CLINICAL TRIAL: NCT02444585
Title: Effect of Denosumab in Reversing Periprosthetic Bone Loss Following Hip Replacement
Brief Title: Longjohn Amgen Study - Effect of Denosumab...
Acronym: EDRPBLFHR
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled in the trial
Sponsor: University of Southern California (Other)
Collaborators: Orthopaedic Institute for Children (Other)
Responsible Party: Principal Investigator, Donald Longjohn, Assistant Professor of Clinical Orthopaedics, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HS-14-00135
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Arthroplasty, Replacement, Hip
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): Drug for prevention of bone loss
  Interventions: Drug: Denosumab
- Control (Placebo Comparator): Hip Replacement Patient without Drug
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Intended to prevent periprosthetic loss of bone mineral density
  Other Names: Prolia

SUMMARY:
The overall objective of the proposed study is to quantify bone loss around non-cemented total hip replacement femoral and acetabular components using DEXA analysis in patients receiving Prolia (denosumab) in the first year of follow up after total hip joint replacement surgery, and to compare this to bone loss in control hip replacement patients receiving a placebo.

The primary outcome variable will be the difference in loss of bone mineral density between the experimental group taking denosumab and the placebo control group, calculated as a percentage, in Gruen Zone 7, the proximal medial calcar region of the femur, over a follow-up period of 12 post-operative months.

The secondary objectives will be to assess the following variables:

* Bone turnover differences between the experimental group taking denosumab and the placebo control group, utilizing serum C-terminal cross-linking telopeptides of type I collagen (CTX-I) (bone resorption) and N-terminal propeptides of type I procollagen (P1NP) (bone formation).
* Difference in loss of bone mineral density between the experimental group taking denosumab and the placebo control group, calculated as a percentage, in each of Gruen Zones 1 through 6, periprosthetic femur.
* Difference in loss of bone mineral density between the experimental group taking denosumab and the placebo control group, calculated as a percentage, in each of DeLee and Charnley's Zones 1 through 3, periprosthetic acetabulum.

Exploratory objectives will be to assess difference in loss of bone mineral density in the contralateral, or non-operated femur for both experimental and control groups, and to determine the role that covariates such as weight, gender, age, baseline BMD, and implant type have on percent change in BMD at 12 months.

DETAILED DESCRIPTION:
EXPERIMENTAL PLAN Study Design The proposed study is a Phase 3, double-blinded, randomized controlled study. All of the 80 patients, both placebo and denosumab groups, will adhere to the same protocol. Patient screening will be performed by the orthopaedic surgeons (Donald Longjohn, MD and Daniel Oakes, MD) during the preoperative clinical appointments, based on the Inclusion and Exclusion Criteria. If the patient is deemed appropriate for the study, consent for participation in the proposed study will be obtained prior to hip replacement surgery.

Two doses of denosumab will be given, 60 mg each. Study Day 1 will be defined as the day of injection, with the first 60 mg dose of denosumab or the placebo administered within 7-14 days following hip replacement surgery. The second injection (60 mg) of either denosumab or the placebo will be administered 6 months after Study Visit #1 . DEXA will be performed on the treated femur using the 7 Gruen radiographic zones of interest, and on the contralateral femur, using traditional analysis protocol, as well as the acetabulum on the treated side using the 3 zones of interest . This will be performed at (1) Study Visit #1, date of first injection; (2) 3 months after injection; (3) 6 months after injection, immediately prior to injection #2; and (4) 12 months after Study Visit #1. Bone mineral density in all patients will be assessed utilizing a Hologic Bone Densitometer with software for metal subtraction on the treated femur. As well, bone turnover markers will be determined base line from blood drawn: (1) at Study Visit #1, date of first injection; (2) 1 month after injection; (3) 3 months after injection; (4) 6 months after injection 1, date of injection 2; (5) 12 months after injection #1 (same as 6 months after injection 2).

Number of Centers

(1) - Orthopaedic Institute for Children (Orthopaedic Hospital), 403 W. Adams Boulevard, Los Angeles, CA

Number of Subjects Number of Subjects = 80

Estimated Study Duration Twenty four (24) months. The study duration for individual participants will be twelve (12) months: Enrollment will take place over the course of the first 12 months of the study and each patient will be followed for 12 months following joint replacement surgery, for a total duration of 24 months. If the study enrollment is not complete by the end of the first 12 months, the enrollment period will be extended an additional 6 months.

SUBJECT ELIGIBILITY Inclusion Criteria Inclusion criteria will allocate patients undergoing elective total hip replacement due to osteoarthritis. The prosthetic device will be a standard, non-cemented tapered total hip replacement, such as an Alloclassic® (Zimmer, Inc., Warsaw, IN) or a similarly shaped implant of the same material (titanium alloy) such as the Summit Hip (Depuy, Inc., Warsaw, IN). Subjects will be between 55 and 75 years of age. Both genders will be included. Prior to surgery, creatinine clearance, calcium, and vitamin D will be checked. Creatinine clearance rates must be above 30 ml/min, vitamin D serum levels must be greater than 12 ng/ml, and patients cannot be hypocalcemic. If vitamin D serum levels are below normal (30ng/ml) the 1000 mg of calcium and at least 1000 Units of vitamin D, recommended by the surgeon at the time of operation will likely be sufficient to correct this problem.

Exclusion Criteria Current use of medications that may affect bone and mineral metabolism (e.g., glucocorticoids, diuretics, estrogen, oral contraceptives, tamoxifen, bisphosphonates, raloxifene, calcitonin, PTH, anticonvulsants, immunosuppressants), and subjects with a history of any disease that affects bone and mineral metabolism (e.g., thyrotoxicosis, hyperparathyroidism, hypocalcemia hypoparathyroidism, chronic renal failure, Cushing's disease, rheumatoid arthritis, hematological disease, alcohol abuse > 3 drinks a day), cancer. Additionally, patients who are taking immunosuppressants will be excluded. Patients who have been treated with anti-TNF in the past 3 months will be excluded. Patients with hypocalcemia or patients who have used bisphosphonates in the 2-3 years prior to the surgery will be excluded. Additionally, patients with creatinine clearance rates below 30 ml/minwill be excluded, as will patients with severe vitamin D deficiencies (<12 ng/ml). Patients with decreased hepatic function as measured by AST, ALT, Alkaline Phosphatase or Total Bilirubin will be excluded from the study. Patients who have had any solid organ or bone marrow transplants will be excluded. Patients who have a history of malignancy within the past 5 years, with the exception of basal cell carcinoma or cervical carcinoma in situ, will be excluded. Additionally, as the incidence of serious infections may be higher in patients treated with denosumab, patients with poorly controlled diabetes/HbA1C will be excluded.

SUBJECT ENROLLMENT AND TREATMENT ASSIGNMENT A total of 80 subjects (N=80) will be enrolled over the first twelve months of the proposed study.

40 of the patients will randomly receive the placebo treatment, and 40 will receive the denosumab treatment. All individuals interacting with patients, including operating surgeons and the patients, will be blinded, with the exception of the Orthopaedic Hospital pharmacist who will be un-blinded. The pharmacist will be in charge of receiving and maintaining the drug until the time of administering to the patient.

TREATMENT PROCEDURES Amgen Investigational Product Denosumab

Dosage, Administration, and Schedule On postoperative day 7-14 (Study Visit #1), and at 6 months following Study Visit #1 (date of first injection, DEXA, and blood draw), the patients will receive either 60 mg denosumab or placebo.

Dose Escalation and Stopping Rules There will be no dose escalation. Therapy will be evaluated if the subject develops symptomatic hypocalcemia, serious skin infections, osteonecrosis of the jaw, or pancreatitis. The subjects will be advised to seek prompt medical attention if they develop any of these signs or symptoms. If Adverse Events develop as defined in section 9.1., if there is suspicion that it may be related to the drug, the case(s) will be investigated and, if deemed necessary, then the patient and doctors may be un-blinded for the purposes of treatment. If symptoms develop after Study Visit #6 (date of second and final injection), even if un-blinding occurs for treatment purposes, patient will be asked to come back for final Study Visit (#5) for 12 month DEXA and blood draw, if willing. If serious side effects occur prior to second injection (Study Visit #4), patient may not receive second injection if there are serious medical concerns.

Dosage Adjustments There will be no dose adjustments.

Concomitant Therapy Subjects will be instructed to take 1000 mg of calcium and at least 1000 Units of vitamin D per day.

Prescribed Therapy during Study Period No use of the medications as listed in the exclusion criteria.

Other Treatment Procedures None

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will allocate patients undergoing elective total hip replacement due to osteoarthritis. The prosthetic device will be a standard, non-cemented tapered total hip replacement, such as an Alloclassic® (Zimmer, Inc., Warsaw, IN) or a similarly shaped implant of the same material (titanium alloy) such as the Summit Hip (Depuy, Inc., Warsaw, IN). Subjects will be between 55 and 75 years of age. Both genders will be included. Prior to surgery, creatinine clearance, calcium, and vitamin D will be checked. Creatinine clearance rates must be above 30 ml/min, vitamin D serum levels must be greater than 12 ng/ml, and patients cannot be hypocalcemic. If vitamin D serum levels are below normal (30ng/ml) the 1000 mg of calcium and at least 1000 Units of vitamin D, recommended by the surgeon at the time of operation will likely be sufficient to correct this problem.

Exclusion Criteria:

* Current use of medications that may affect bone and mineral metabolism (e.g., glucocorticoids, diuretics, estrogen, oral contraceptives, tamoxifen, bisphosphonates, raloxifene, calcitonin, PTH, anticonvulsants, immunosuppressants), and subjects with a history of any disease that affects bone and mineral metabolism (e.g., thyrotoxicosis, hyperparathyroidism, hypocalcemia hypoparathyroidism, chronic renal failure, Cushing's disease, rheumatoid arthritis, hematological disease, alcohol abuse > 3 drinks a day), cancer. Additionally, patients who are taking immunosuppressants will be excluded. Patients who have been treated with anti-TNF in the past 3 months will be excluded. Patients with hypocalcemia or patients who have used bisphosphonates in the 2-3 years prior to the surgery will be excluded. Additionally, patients with creatinine clearance rates below 30 ml/minwill be excluded, as will patients with severe vitamin D deficiencies (<12 ng/ml). Patients with decreased hepatic function as measured by AST, ALT, Alkaline Phosphatase or Total Bilirubin will be excluded from the study. Patients who have had any solid organ or bone marrow transplants will be excluded. Patients who have a history of malignancy within the past 5 years, with the exception of basal cell carcinoma or cervical carcinoma in situ, will be excluded. Additionally, as the incidence of serious infections may be higher in patients treated with denosumab, patients with poorly controlled diabetes/HbA1C will be excluded.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Bone Mineral Density | One Year
  The primary outcome variable will be the difference in loss of bone mineral density between the experimental group taking denosumab and the placebo control group.

SECONDARY OUTCOMES:
Bone Turnover Markers | One Year
  Bone turnover differences between the experimental group taking denosumab and the placebo control group.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Longjohn, MD, Principal Investigator — University of Southern California; Edward Ebramzadeh, PhD, Study Director — Orthopaedic Institute for Children (Orthopaedic Hospital)
Locations (1):
- Keck Medicine of USC, Los Angeles, California, United States